CLINICAL TRIAL: NCT00421629
Title: Experimental Study to Assess Interventions Aimed at Improving the Equity Impact of Community-Based Health Insurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: PHHPBD25; GR067926MA
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2007-01

CONDITIONS: Health Insurance
Keywords: health insurance; hospitalization insurance; community based health insurance; health care access; developing countries; randomized controlled trials
MeSH Terms: interventions — Prospective Payment System

INTERVENTIONS:
Behavioral: After-sales service and supportive supervision (AfterSS)
Behavioral: Prospective reimbursement (PR)
Behavioral: Both (AfterSS and PR)

SUMMARY:
The purpose of this study is to assesses interventions aimed at improving the distributional impact of a community based health insurance scheme in rural India.

DETAILED DESCRIPTION:
Community based health insurance is often cited as a means of improving access and financial protection in developing countries, but such schemes may not benefit the poorest. We evaluate alternative strategies for improving the uptake of benefits of a community based health insurance scheme by its poorest members.

Comparisons: Three groups are compared to standard insurance scheme members (Control). One group is provided with after-sale service and supportive supervision (AfterSS). A second group is provided with prospective reimbursement (PR). A third group is provided with these two interventions together (Both).

ELIGIBILITY:
Subdistrict Inclusion Criteria:

* 500 or more female (>=18 y of age) SEWA Insurance members in 2003

Subdistrict Exclusion Criteria:

* All members were mandatorily enrolled in the scheme by a donor agency
* Ahe sub-district had no general hospital of 25 beds or more

Individual Inclusion Criteria:

* All female and male members of SEWA Insurance for 2004 and 2005

Individual Exclusion Criteria:

* Those whose home could not be found based on given address data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 688
Dates: Start 2003-10; Study Completion 2006-04

PRIMARY OUTCOMES:
socioeconomic status of claimants relative to the membership base in their subdistricts of residence

SECONDARY OUTCOMES:
enrolment rates in Vimo SEWA
mean socioeconomic of the insured relative to the general rural population
rate of insurance claim submission

CONTACTS AND LOCATIONS:
Overall Officials: Anne J Mills, MA DHSA PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Michael K Ranson, MD MPH PHD, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- Self Employed Women's Association, Ahmedabad, Gujarat, India

REFERENCES:
- [Background] Ranson MK, Sinha T, Chatterjee M, Acharya A, Bhavsar A, Morris SS, Mills AJ. Making health insurance work for the poor: learning from the Self-Employed Women's Association's (SEWA) community-based health insurance scheme in India. Soc Sci Med. 2006 Feb;62(3):707-20. doi: 10.1016/j.socscimed.2005.06.037. Epub 2005 Jul 28. PMID 16054740
- [Background] Sinha T, Ranson MK, Chatterjee M, Acharya A, Mills AJ. Barriers to accessing benefits in a community-based insurance scheme: lessons learnt from SEWA Insurance, Gujarat. Health Policy Plan. 2006 Mar;21(2):132-42. doi: 10.1093/heapol/czj010. Epub 2005 Dec 22. PMID 16373360
- [Background] Ranson MK, Sinha T, Morris SS, Mills AJ. CRTs--cluster randomized trials or "courting real troubles": challenges of running a CRT in rural Gujarat, India. Can J Public Health. 2006 Jan-Feb;97(1):72-5. doi: 10.1007/BF03405220. PMID 16512334
- [Background] Morris SS, Ranson MK, Sinha T, Mills AJ. Measuring improved targeting of health interventions to the poor in the context of a community-randomised trial in rural India. Contemp Clin Trials. 2007 Jul;28(4):382-90. doi: 10.1016/j.cct.2006.10.008. Epub 2006 Oct 14. PMID 17126613
- [Background] Ranson MK, Sinha T, Gandhi F, Jayswal R, Mills AJ. Helping members of a community-based health insurance scheme access quality inpatient care through development of a preferred provider system in rural Gujarat. Natl Med J India. 2006 Sep-Oct;19(5):274-82. PMID 17203684